CLINICAL TRIAL: NCT01359020
Title: Randomized, Open Label, Comparative, Parallel, Multicenter Trial to Determinate the Efficacy Anf Tolerability of Ibuprofen, Acetaminophen and Dipyrone Drops to Fever Control in Children
Brief Title: Ibuprofen, Acetaminophen and Dipyrone to Fever Control in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mantecorp Industria Quimica e Farmaceutica Ltd. (Industry)
Responsible Party: Claudia Domingues, Mantecorp
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALI/P/04-1
Record Dates: First submitted 2011-05-20; First posted 2011-05-24 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2011-05

CONDITIONS: Fever
Keywords: Fever; Ibuprofen; Acetaminophen; Dipyrone
MeSH Terms: conditions — Fever | interventions — Ibuprofen; Dipyrone; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ibuprofen (Experimental): 10 milligram per kilo, oral administration
  Interventions: Drug: ibuprofen, dipyrone, acetaminophen
- Acetaminophen (Active Comparator): 10 milligram per kilo, oral administration
  Interventions: Drug: ibuprofen, dipyrone, acetaminophen
- Dipyrone (Active Comparator): 10 milligram per kilo, oral administration
  Interventions: Drug: ibuprofen, dipyrone, acetaminophen

INTERVENTIONS:
Drug: ibuprofen, dipyrone, acetaminophen — The dosage for the three drugs was the same: 10 milligrams per kilo, oral administration

SUMMARY:
The purpose of this study was to compare the efficacy and tolerability of acetaminophen, dipyrone and ibuprofen to fever control in children.

For the efficacy asses were compared:

* the time to start the action;
* the action duration;
* the difference between the basal temperature and the lower temperature in the study period.

For the tolerability asses all adverse events were recorded, as well as your intensity and the relation to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* male and female children aged 06 months to 06 years old, weight above 5 kilo and axillary temperature above 37,5 celsius degree.

Exclusion Criteria:

* patients with a bad general heath state
* patients with neoplasia, pepic ulcer, gastrointestinal bleeding,history of fever convulsion;
* intolerant to dypirone, ibuprofen, acetaminophen or any other nonsteroidal antiinflammatory drug;
* moderated or severe dehydration;
* conscience state alteration;
* not capable of ingest oral drugs;
* patients being treated with steroids;
* patients treated with antiinflammatory, analgesic and antipyretic drugs in the last 06 hours before the study.

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 396 (Actual)
Dates: Start 2007-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Antipyretic efficacy | Temperature was verified 15, 30, 45 and 60 minutes, 2, 3, 4, 5, 6, 7 and 8 hours after the administration of the drug.
  The antipyretic efficacy was assessed comparing the time to the beggining of the action of the drugs, the difference between the final and inicial temperature and time of action.

SECONDARY OUTCOMES:
Adverse Events | Adverse Events were verified at 15, 30, 45 and 60 minutes, 2, 3, 4, 5, 6, 7 and 8 hours after the administration of the drug.
  All adverse events were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Patrícia DN Moura, Study Director — Mantecorp Indústria Química e Farmacêutica Ltda.
Locations (1):
- Instituto de Medicina Integral Professor Fernando Figueira, Recife, Pernambuco, Brazil